CLINICAL TRIAL: NCT03091829
Title: Chest Pain Unit II Register - CPU II Register
Brief Title: Chest Pain Unit II Register
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: CPU II Register
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2019-09

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicentric, prospective, non-interventional observational study with two parts:

1. A register of quality assurance within the recertification of clinics
2. An extended register with scientific protocol.

DETAILED DESCRIPTION:
1. Quality assurance

   As a quality-assuring basic register, the CPU II register checks the extent to which certified Chest Pain Units fulfill the criteria published by the DGK. In particular, the following quality dimensions are evaluated:
   * Indication quality
   * Diagnostic quality
   * Therapeutic quality
   * Structural quality / networking
2. Platform for projects with a scientific focus

The CPU II register and the infrastructure provided are a platform for further projects with scientific questions (scientific protocol = WP):

WP: Clinical history after CPU (PCI data / discharge / 12-month FUP) in patients with leading cardiac diagnosis

ELIGIBILITY:
Inclusion Criteria:

* CPU patient
* > 18 years
* Written consent of the patient

Exclusion Criteria:

* Denied consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Basic register:
  All patients who are admitted to a CPU.
  Scientific Protocol:
  All patients who are admitted to a CPU and have their consent to participate in a follow-up (in patients with leading cardiac diagnosis).
Sampling Method: Non-Probability Sample
Enrollment: 4829 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Fulfillment of DGK criteria | 12 months
  Quality assurance: Fulfillment of the recertification criteria of the german society for cardiology
Clinical progress after CPU | 12 months
  Scientific protocol: Documentation of the clinical progress after CPU

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Städtisches Klinikum Neuperlach, München, Bavaria
  - Klinikum der Johannes-Gutenberg-Universität, 2. Med. Klinik, Mainz, RLP
  - Klinikum Links der Weser Bremen, Bremen

IPD SHARING:
Plan to Share IPD: No